CLINICAL TRIAL: NCT01214135
Title: A Retrospective, Non-interventional Study to Evaluate the Use of Seroquel XR and Seroquel IR in the Clinical Practice of Inpatients With Schizophrenia
Brief Title: A Retrospective Non-interventional Study to Evaluate the Use of Seroquel Extended Release (XR) and Immediate Release (IR) in the Clinical Practice of Inpatients With Schizophrenia
Acronym: SPIN
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca
Other Study IDs: NIS-NSE-SER-2010/1
Record Dates: First submitted 2010-09-24; First posted 2010-10-04 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Schizophrenia
Keywords: Mental disorder; antipsychotic treatment
MeSH Terms: conditions — Schizophrenia; Mental Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with a diagnosis of schizophrenia who have been hospitalized and received at least one dose of Seroquel XR or Seroquel IR during the study period (1st of July 2009 - 30th of September 2010).

SUMMARY:
The primary objective of this non-interventional study is to investigate how Seroquel XR and Seroquel IR are used in the clinical practice of inpatients with schizophrenia. This will be done by a retrospective review of medical records to evaluate patients treated with Seroquel XR or Seroquel IR as primary antipsychotic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia.
* At least one dose of Seroquel XR or Seroquel IR during the study period (1st of July 2009 - 30th of September 2010).
* Hospitalization due to psychotic symptoms at any time during the study period (1st of July 2009 - 30th of September 2010) and with admission and discharge dates available.

Exclusion Criteria:

* Participation in a clinical trial during the study period.
* Treatment in forensic care according to LRV ("Lagen om Rättspsykiatrisk Vård").

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 300 patients with schizophrenia who have been hospitalized during the study period (1st of July 2009 - 30th of September 2010).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To investigate how Seroquel XR and Seroquel IR are used in the clinical practice of inpatients with schizophrenia | every day for the time period of 15 Oct to 31 Dec 2010

SECONDARY OUTCOMES:
To investigate comorbidities of patients with schizophrenia receiving Seroquel XR and IR | every day for the time period of 15 Oct to 31 Dec 2010
To investigate whether Seroquel XR and Seroquel IR are used to treat different types of inpatients with schizophrenia by evaluation of patient characteristics | every day for the time period of 15 Oct to 31 Dec 2010
To investigate the treatment sequence of Seroquel XR and Seroquel IR in the clinical practice of patients with schizophrenia by evaluation of duration, dosage, reason for treatment, and, if applicable, reason for change, with Seroquel XR and Seroquel IR | every day for the time period of 15 Oct to 31 Dec 2010

CONTACTS AND LOCATIONS:
Overall Officials: Dr Eva Dencker Vansvik, MD, Study Director — AstraZeneca; Dr Lars Eriksson, MD, Principal Investigator — Rättspsykiatriska Vårdkedjan, Hisings-Backa, Sweden
Locations (14):
- Sweden (14):
  - Research Site, Falköping
  - Research Site, Gothenburg
  - Research Site, Helsingborg
  - Research Site, Karlskrona
  - Research Site, Karlstad
  - Research Site, Lund
  - Research Site, Malmo
  - Research Site, Mölndal
  - Research Site, Öjebyn
  - Research Site, Stockholm
  - Research Site, Trollhättan
  - Research Site, Umeå
  - Research Site, Uppsala
  - Research Site, Vaxjo

REFERENCES:
- [Derived] Eriksson L, Hallerback T, Jorgensen L, Carlborg A. Use of quetiapine XR and quetiapine IR in clinical practice for hospitalized patients with schizophrenia: a retrospective study. Ther Adv Psychopharmacol. 2012 Dec;2(6):217-26. doi: 10.1177/2045125312453935. PMID 23983980